CLINICAL TRIAL: NCT00876902
Title: A Controlled, Prospective, Blinded, Randomized, Single-Center, Study of YSPSL for Prevention of Ischemic Reperfusion Injury in Patients Undergoing Cadaveric Orthotopic Liver Transplantation
Brief Title: YSPSL for Prevention of Ischemic Reperfusion Injury in Patients Undergoing Cadaveric Orthotopic Liver Transplantation
Acronym: YSPSL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Y's Therapeutics, Inc. (Industry)
Responsible Party: Stefan Hemmerich, Clinical Operations, Y's Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YSPSL-0003-PF.3; IND 101,040
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Ischemia Reperfusion Injury
Keywords: liver transplantation; cadaveric liver transplantation; ischemic reperfusion injury; primary non-function; delayed non-Function; poor early graft function; YSPSL; recombinant PSGL-Ig
MeSH Terms: conditions — Reperfusion Injury | interventions — University of Wisconsin-lactobionate solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active Group: (18 subjects) YSPSL administered as an ex vivo flush (20 mg YSPSL in Viaspan® 200 mL total volume) into the portal vein prior to transplant at the back table; YSPSL 1 mg/kg administered IV to the transplant recipient PRIOR to arterial reperfusion of the liver. One extra IV dose of 1 mg/kg will be given at the end of the procedure only to patients that have experienced an intraoperative blood loss of greater than 10 units.
  Interventions: Drug: recombinant P-selectin glycoprotein ligand Ig fusion protein
- 2 (Placebo Comparator): Placebo Control: (18 subjects) Ex vivo flush of placebo control (200 mL Viaspan®) into the portal vein prior to transplant and 0.1 mL/kg placebo control (saline) IV to the transplant recipient PRIOR to arterial reperfusion of the liver. One additional infusion of 0.1 mL/kg placebo control (saline) will be given at the end of the procedure to patients that have experienced an intraoperative blood loss of greater than 10 units.
  Interventions: Drug: Viaspan® and saline

INTERVENTIONS:
Drug: recombinant P-selectin glycoprotein ligand Ig fusion protein — The active study drug dose includes both a 1 mg/kg IV infusion for the recipient and a 20 mg [approximately 0.27 mg/kg] as an ex vivo flush. The doses will be administered via 2 separate infusions of study agent: one 20 mg dose into the portal vein of the liver prior to implantation as an ex vivo flush with Viaspan®; and the second infusion of 1 mg/kg intravenously into the recipient, when technically feasible, prior to the hepatic artery anastomosis. Those patients that experience an intraoperative blood loss of >10 units, will receive an additional 1 mg/kg IV infusion of study agent at the end of the transplant surgery.
  Other Names: rPSGL-Ig; Torapsel
  Arms: 1
Drug: Viaspan® and saline — Placebo of a volume equivalent to active study drug will be prepared for administration to the control group to help maintain the blind. Those patients that experience an intraoperative blood loss of >10 units, will receive an additional 1 mg/kg IV infusion of placebo equivalent at the end of the transplant surgery.
  Other Names: Placebo
  Arms: 2

SUMMARY:
The study is designed to assess the feasibility of evaluating YSPSL for the amelioration of ischemia reperfusion injury following liver transplantation by administering YSPSL into the liver graft directly ex vivo via the portal vein and to the recipient intravenously prior to reperfusion. This study is an extension of the recent pilot study YSPSL-0002 with an almost identical study protocol. The rationale of this and the previous study is based on the recent observation that P-selectin expression has been associated in liver grafts with prolonged cold storage times and rejection. By examining biomarkers of IRI including P-selectin by immunohistochemistry and/or quantitative PCR, liver histology and hepatic blood flow using established techniques, the goal of this study is to evaluate the feasibility of using these modalities for future studies of safety and efficacy.

DETAILED DESCRIPTION:
YSPSL-0003 is an extension into 36 patients of the previous 12 patient pilot study YSPSL-0002 under an almost identical study protocol with extended inclusion criteria. Like YSPSL-0002, YSPSL-0003 is a single-center (UCLA), randomized, placebo-controlled, double-blind study. Patients are randomly assigned to either active study drug (Active group) or placebo (Control group) prior to transplantation. The active study drug dose includes both a 1 mg/kg IV infusion for the recipient and a 20 mg [approximately 0.27 mg/kg] as an ex vivo flush. The doses are administered via 2 separate infusions of study agent: one 20 mg dose into the portal vein of the liver prior to implantation as an ex vivo flush with Viaspan®; and the second infusion of 1 mg/kg intravenously into the recipient, when technically feasible, prior to the hepatic artery anastomosis. Placebo of a volume equivalent to active study drug is prepared for administration to the control group to help maintain the blind. Those patients that experience an intraoperative blood loss of >10 units, receive an additional 1 mg/kg IV infusion of study agent (or placebo equivalent) at the end of the transplant surgery. The Investigator/Sponsor is blinded to the treatment assignment for each patient. Randomization assignment is maintained by UCLA's clinical pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be a recipient of a primary (first) ABO compatible cadaveric liver allograft
* Patient's age is less than 18 years
* Patient is not a recipient of a multivisceral transplant or simultaneous kidney transplant
* Patient has not undergone prior organ or cellular transplant of any type
* Patient has a Model for End Stage Liver Disease (MELD) score of ≤38
* Cold ischemia time (CIT) anticipated to be less than 14 hours
* Donor liver procured by UCLA liver team
* Veno-veno bypass is not planned to be used for the patient (e.g. no prior surgery or other factor that indicates a risk for excessive blood loss and therefore a need for veno-veno bypass +/- autologous recovery during surgery)
* For patients who are women of childbearing potential, patient has a negative pregnancy test (either urine or serum) within 48 hours prior to transplant
* Patient (male and female) is willing to use an acceptable form of birth control for at least 3 months post-treatment
* Patient is willing and able to sign informed consent.

Exclusion Criteria:

* Patient has a prior organ transplant of any type
* Patient has known allergic or intolerance reactions to human immune globulins, antibodies, or components of the formulation or known contraindication to administration of YSPSL
* Patient has an uncontrolled active infection (on antibiotics with controlled infection is not an exclusion)
* Patient has active Hepatitis B virus (HBV)/transplant for HBV related cirrhosis
* Patient has previously participated in this study or another study with YSPSL
* Patient has received investigational therapy within 90 days prior to the transplant procedure
* Patient has current drug or alcohol abuse or, in the opinion of the investigator, is at risk for poor compliance with the visits in this protocol (no drug testing required)
* Patient is a pregnant or nursing female, a female of childbearing potential planning to become pregnant within the duration of this study, or is not practicing birth control
* Patient is planned to receive a living donor liver transplant
* Patient lives >200 miles away or otherwise is not able to participate in study follow-up visits
* Donor body mass index >40
* Donor liver biopsy >40% macrosteatotic fat
* Donor age >70.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Safety will be evaluated by clinical and laboratory assessments, an abbreviated pharmacokinetic (PK) profile of the administered dose of YSPSL, and graft function and patient and graft survival through 6 months post-transplant. | 6 months post trasplant

SECONDARY OUTCOMES:
To evaluate the potential efficacy of prophylaxis with YSPSL on ischemia reperfusion injury (IRI) as assessed by proposed efficacy evaluations of IRI in liver transplants, in patients who meet eligibility criteria for the trial. | 6 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hemmerich, PhD, Study Director — Y's Therapeutics, Inc.
Locations (1):
- UCLA School of Medicine, Los Angeles, California, United States

REFERENCES:
- [Background] Amersi F, Farmer DG, Shaw GD, Kato H, Coito AJ, Kaldas F, Zhao D, Lassman CR, Melinek J, Ma J, Volk HD, Kupiec-Weglinski JW, Busuttil RW. P-selectin glycoprotein ligand-1 (rPSGL-Ig)-mediated blockade of CD62 selectin molecules protects rat steatotic liver grafts from ischemia/reperfusion injury. Am J Transplant. 2002 Aug;2(7):600-8. doi: 10.1034/j.1600-6143.2002.20704.x. PMID 12201360
- [Derived] Busuttil RW, Lipshutz GS, Kupiec-Weglinski JW, Ponthieux S, Gjertson DW, Cheadle C, Watkins T, Ehrlich E, Katz E, Squiers EC, Rabb H, Hemmerich S. rPSGL-Ig for improvement of early liver allograft function: a double-blind, placebo-controlled, single-center phase II study. Am J Transplant. 2011 Apr;11(4):786-97. doi: 10.1111/j.1600-6143.2011.03441.x. Epub 2011 Mar 14. PMID 21401865
- See also: YSPSL (rPSGL-Ig) treatment affords benefit in animal model of liver transplantation — http://www.ncbi.nlm.nih.gov/pubmed/12201360?ordinalpos=2&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum